CLINICAL TRIAL: NCT02838511
Title: Which is a Better Measure of Frailty in Perioperative Setting: Deficit Accumulation Model or Phenotype Model?
Brief Title: Measure of Frailty in Perioperative Setting
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1241
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-cardiac surgery: Hopkins Frailty Score (HFS) or Modified Frailty Index (MFI) will be obtained during during pre anesthesia evaluation
  Interventions: Other: Modified Frailty Index (MFI); Other: Hopkins Frailty Score (HFS)

INTERVENTIONS:
Other: Modified Frailty Index (MFI) — non-cardiac surgical patients will have frailty evaluated
Other: Hopkins Frailty Score (HFS) — non-cardiac surgical patients will have frailty evaluated

SUMMARY:
Though most physicians believe they can identify frail patients, frailty is a poorly characterized and complex clinical syndrome. Frailty has been categorized four dimensions by de Vries et al: 1) physical (physical activity, nutrition, mobility, strength and energy); 2) biochemical (nutritional and inflammatory biomarkers); 3) psychological (cognition and mood); and, 4) social (social contact and support). 1 However, the pathophysiology of frailty remains unclear. Two broad hypotheses have been proposed.

Deficit accumulation model: This hypothesis assumes that frailty occurs due to accumulation and additive effect of multiple deficits, which occur across various domains. The more deficits a person has, the more likely that person is to be frail. Frailty in this paradigm is thus measured by identifying the number of positive factors/ deficits from a list. This is used to create a proportional index of deficits, expressed as the ratio of deficits present to the total number of deficits considered.

Many studies have used a modified frailty index (MFI) with 11 factors, which has shown to correlate well with patient outcomes after surgery.

Phenotype model: Fried et al in 2001 proposed a phenotype based model, in which she identified various clinical features that define frailty as a clinical syndrome. This criterion, known as Fried index, consists of 5 factors- shrinking, weakness, exhaustion, slowness, and low physical activity level. The Fried index is the most commonly used phenotype-based assessment tool to evaluate frailty. An advantage is its ease-of use during preoperative visits. Measurement of these factors in a perioperative setting was further characterized by Makary et al in 2010, and was the basis for the Hopkins Frailty Score (HFS).

Currently, there exists no gold standard for assessment of frailty, especially in the perioperative setting. In the absence of a well-accepted gold standard, a measurement of frailty which would predict adverse postoperative outcomes would be useful. However, no study has compared the prognostic abilities of HFS and MFI, after non-cardiac surgery.

All adult patients presenting to pre anesthesia evaluation clinic (PACE) at Cleveland Clinic main campus will be included in the this prospective observational cohort study. Frailty would be evaluated prospectively using HFS and components of MFI will be obtained from Cleveland Clinic Perioperative Health Documentation System registry (PHDS).

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18-100 years of age)
* patients presenting to the PACE clinic for non cardiac surgery

Exclusion Criteria:

* children (under 18 years of age)
* patients presenting to the PACE clinic for cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to pre anesthesia evaluation clinic at Cleveland clinic main campus.
Sampling Method: Probability Sample
Enrollment: 1190 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Days in Hospital | 30 days after non-cardiac surgery
  total number of days spent by patient in the hospital within 30 days of non-cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No